CLINICAL TRIAL: NCT03588286
Title: Programmed Ventricular Stimulation to Risk Stratify for Early Cardioverter-Defibrillator (ICD) Implantation to Prevent Tachyarrhythmias Following Acute Myocardial Infarction (PROTECT-ICD)
Acronym: PROTECT-ICD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Pramesh Kovoor, Senior Staff Specialist Cardiologist, Western Sydney Local Health District
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PROTECT-ICD, Version 5; ACTRN12614000042640 (Registry Identifier: ANZCTR)
Record Dates: First submitted 2018-07-04; First posted 2018-07-17 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Sudden Cardiac Death
Keywords: Myocardial Infarction (MI), Sudden Cardiac Death (SCD), Electrophysiological Study (EPS), Ventricular Tachycardia (VT)
MeSH Terms: conditions — Death, Sudden, Cardiac; Myocardial Infarction; Tachycardia, Ventricular | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Early EPS) (Experimental): The intervention group all undergo electrophysiologic study early after myocardial infarction (within 40 days of MI).
  If the study is positive (inducible monomorphic ventricular tachycardia of cycle length greater than or equal to 200ms) participants have an ICD implanted. Participants with a negative study (no inducible arrhythmia or induced ventricular fibrillation/ ventricular flutter cycle length <200ms) are discharged without an ICD.
  A proportion of trial patients from both the intervention and control arms at >48 hours following revascularisation for STEMI will undergo CMR to enable correlation with (1) inducible VT at EPS and (2) SCD and non-fatal arrhythmia on follow up. CMR will simultaneously assess left ventricular function, ventricular strain, myocardial infarction size, and peri-infarction injury.
  Interventions: Procedure: Electrophysiology study (EPS); Procedure: Cardiac Magnetic Resonance (CMR)
- Control Arm (Standard Care) (Active Comparator): The control group receive ongoing standard care according to the practise of their institution. This includes discharge from hospital as per their treating physician and follow up as usual in the community. Participants in this group would be eligible to receive an ICD according to the standard practise of their cardiologist (guideline recommendations are after 40 days following myocardial infarction or 90 days following revascularisation only in patients with left ventricular ejection fraction less than or equal to 30% or less than or equal to 35% in the presence of heart failure).
  A proportion of trial patients from both the intervention and control arms at >48 hours following revascularisation for STEMI will undergo CMR to enable correlation with (1) inducible VT at EPS and (2) SCD and non-fatal arrhythmia on follow up. CMR will simultaneously assess left ventricular function, ventricular strain, myocardial infarction size, and peri-infarction injury.
  Interventions: Other: Standard Care; Procedure: Cardiac Magnetic Resonance (CMR)

INTERVENTIONS:
Procedure: Electrophysiology study (EPS) — EPS will be performed in all patients in the intervention arm with programmed ventricular stimulation with a drive train of 8 beats at 400 ms with up to 4 extrastimuli and stimulation from the right ventricular apex with current delivered at twice pacing threshold. The end point for stimulation will be sustained monomorphic ventricular tachycardia (VT) lasting > 10 seconds. If sustained monomorphic VT with cycle length (CL) ≥200ms is induced by ≤4 extra stimuli the EPS result will be considered positive for inducible VT.30 Ventricular fibrillation or flutter with CL<200ms will be considered a negative result. The Programmed Ventricular Stimulation (PVS) induction will be repeated a second time if the initial induction was negative for VT.
  Arms: Intervention Arm (Early EPS)
Other: Standard Care — The control group receive ongoing standard care according to the practise of their institution. This includes discharge from hospital as per their treating physician and follow up as usual in the community. Participants in this group would be eligible to receive an ICD according to the standard practise of their cardiologist (guideline recommendations are after 40 days following myocardial infarction or 90 days following revascularisation only in patients with left ventricular ejection fraction less than or equal to 30% or less than or equal to 35% in the presence of heart failure).
  Arms: Control Arm (Standard Care)
Procedure: Cardiac Magnetic Resonance (CMR) — CMR will be performed on either a 1.5-T or 3-T scanner. Gadolinium contrast (Gd-BOPTA, MultihanceTM) will be administered for quantification myocardial perfusion imaging with subsequent late gadolinium enhanced imaging after a total dose of 0.1mmol/kg. Exclusion criteria specific for CMR will include pregnancy, renal insufficiency defined as glomerular filtration rate (GFR) <30 mL/min, contraindication to MRI (including non-MRI compatible pacemaker/ICD or metal implants, non-MR safe prosthetic heart valves), claustrophobia which cannot be controlled via standard methods (benzodiazepines and/or sedative antihistamine administration) and prior allergic reaction to gadolinium-based contrast agent.

SUMMARY:
The PROTECT-ICD trial is a physician-led, multi-centre randomised controlled trial targeting prevention of sudden cardiac death in patients who have poor cardiac function following a myocardial infarct (MI). The trial aims to assess the role of electrophysiology study (EPS) in guiding implantable cardioverter-defibrillator (ICD) implantation, in patients early following MI (first 40 days). The secondary aim is to assess the utility of cardiac MRI (CMR) in analysing cardiac function and viability as well as predicting inducible and spontaneous ventricular tachyarrhythmia when performed early post MI.

Following a MI patients are at high risk of sudden cardiac death (SCD). The risk is highest in the first 40 days; however, current guidelines exclude patients from receiving an ICD during this time. This limitation is based largely on a single study, The Defibrillator in Acute Myocardial Infarction Trial (DINAMIT), which failed to demonstrate a benefit of early ICD implantation. However, this study was underpowered and used non-invasive tests to identify patients at high risk. EPS identifies patients with the substrate for re-entrant tachyarrhythmia, and has been found in multiple studies to predict patients at risk of SCD. Contrast-enhanced CMR is a non-invasive test without radiation exposure which can be used to assess left ventricular function. In addition, it provides information on myocardial viability, scar size and tissue heterogeneity. It has an emerging role as a predictor of mortality and spontaneous ventricular arrhythmia in patients with a previous MI.

A total of 1,058 patients who are at high risk of SCD based on poor cardiac function (left ventricular ejection fraction (LVEF) ≤40%) following a ST-elevation or non-STE myocardial infarct will be enrolled in the trial. Patients will be randomised 1:1 to either the intervention or control arm.

In the intervention arm all patients undergo early EPS. Patients with a positive study (inducible ventricular tachycardia cycle length ≥200ms) receive an ICD, while patients with a negative study (inducible ventricular fibrillation or no inducible VT) are discharged without an ICD, regardless of the LVEF.

In the control arm patients are treated according to standard local practice. This involves early discharge and repeat assessment of cardiac function after 40 days or after 90 days following revascularisation (PCI or CABG). ICD implantation after 40 days according to current guidelines (LVEF≤30%, or ≤35% with New York Heart Association (NYHA) class II/III symptoms) could be considered, if part of local standard practice, however the ICD is not funded by the trial.

A proportion of trial patients from both the intervention and control arms at >48 hours following MI will undergo CMR to enable correlation with (1) inducible VT at EPS and (2) SCD and non-fatal arrhythmia on follow up. It will be used to simultaneously assess left ventricular function, ventricular strain, myocardial infarction size, and peri-infarction injury. The size of the infarct core, infarct gray zone (as a measure of tissue heterogeneity) and total infarct size will be quantified for each patient.

All patients will be followed for 2 years with a combined primary endpoint of non-fatal arrhythmia and SCD. Non-fatal arrhythmia includes resuscitated cardiac arrest, sustained ventricular tachycardia (VT) and ventricular fibrillation (VF) in participants without an ICD. Secondary endpoints will include all-cause mortality, non-sudden cardiovascular death, non-fatal repeat MI, heart failure and inappropriate ICD denial. Secondary endpoints for CMR correlation will include (1) the presence or absence of inducible VT at EP study, and (2) combined endpoint of appropriate ICD activation or SCD at follow up.

It is anticipated that the intervention arm will reduce the primary endpoint as a result of prevention of a) early sudden cardiac deaths/cardiac arrest, and b) sudden cardiac death/cardiac arrest in patients with a LVEF of 31-40%. It is expected that the 2-year primary endpoint rate will be reduced from 6.7% in the control arm to 2.8% in the intervention arm with a relative risk reduction (RRR) of 68%. A two-group chi-squared test with a 0.05 two-sided significance level will have 80% power to detect the difference between a Group 1 proportion of 0.028 experiencing the primary endpoint and a Group 2 proportion of 0.067 experiencing the primary endpoint when the sample size in each group is 470. Assuming 1% crossover and 10% loss to follow up the required sample size is 1,058 (n=529 patients per arm). To test the hypothesis that tissue heterogeneity at CMR predicts both inducible and spontaneous ventricular tachyarrhythmias will require a sample size of 400 patients to undergo CMR.

It is anticipated that the use of EPS will select a group of patients who will benefit from an ICD soon after a MI. This has the potential to change clinical guidelines and save a large number of lives.

ELIGIBILITY:
Inclusion Criteria:

* 2-40 days (inclusive) following a myocardial infarct
* Impaired left ventricular systolic function (LVEF≤40% or at least moderately impaired)

Exclusion Criteria:

1. Age <18 or >85;
2. Pregnancy;
3. Nursing home resident dependent on one or more activities of daily living;
4. Significant non-cardiac co-morbidity with high likelihood of death within 1 year (this would include any metastatic malignancy, or other terminal disease);
5. Significant psychiatric illnesses that may be aggravated by device implantation or that may preclude regular follow up;
6. Intravenous drug abuse (ongoing);
7. Unresolved infection associated with risk for hematogenous seeding;
8. Pre-existing implantable cardioverter-defibrillator (ICD);
9. Secondary prevention indication for an ICD (i.e. sustained ventricular arrhythmias occurring more than 48 hours after qualifying myocardial infarction (patients with ventricular arrhythmias occurring ≤48 hours of myocardial infarction, or with non-sustained ventricular tachycardia at any time, are not excluded));
10. On the heart transplant list;
11. Recurrent unstable angina despite revascularisation (defined as ongoing chest pain or ischemic symptoms at rest or with minimal exertion despite adequate treatment with anti-anginal medications);**
12. Congestive heart failure New York Heart Association class IV, defined as shortness of breath at rest, which is refractory to medical treatment (not responding to treatment)** **NOTE: patients who meet exclusion based on (11) or (12) can be reviewed again in 2-3 days and if symptoms have resolved or treatment performed can be re-considered for inclusion.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1058 (Estimated)
Dates: Start 2014-02-27 (Actual); Primary Completion 2027-12-06 (Estimated); Study Completion 2029-12-06 (Estimated)

PRIMARY OUTCOMES:
Sudden cardiac death | 2 years after randomisation
  Cause of death will be determined based on information obtained from witnesses, family members, death certificates, hospital records and autopsy or coroner reports. Sudden cardiac death will be explicitly defined as death that occurs "suddenly and unexpectedly" in a patient in otherwise stable condition and includes witnessed instantaneous deaths (with or without documentation of arrhythmia), unwitnessed deaths if the patient had been seen within 24 hours before death (in the absence of another clear cause of death), deaths caused by incessant ventricular tachyarrhythmia, deaths considered a sequel of cardiac arrest and deaths resulting from pro-arrhythmia of anti-arrhythmic drugs.31 The remainder of deaths will be classified as either non-sudden cardiovascular death, or non-cardiovascular death. Operative deaths associated with the implantation of an ICD will be counted as non-sudden cardiovascular death.
Non-fatal arrhythmia | 2 years after randomisation
  Non-fatal arrhythmia includes resuscitated cardiac arrest, sustained ventricular tachycardia (VT) and ventricular fibrillation (VF) in participants without an ICD. Resuscitated cardiac arrest is defined as a sudden circulatory arrest requiring cardiopulmonary resuscitation (CPR) (with or without documented arrhythmia) from which the patient regains consciousness. VT and VF are defined as ECG or telemetry-documented ventricular tachycardia or ventricular fibrillation. Only sustained ventricular tachycardia will be included (greater than 30 seconds of VT) or if the VT required emergency treatment with anti-arrhythmic medications or electrical cardioversion.

SECONDARY OUTCOMES:
All-cause mortality | 2 years after randomisation
  All deaths.
Non-sudden cardiovascular death | 2 years after randomisation
  Non-sudden cardiovascular deaths will be classified as death due to myocardial infarction, heart failure or another cardiovascular cause including cerebrovascular or peripheral vascular causes.
Non-fatal repeat MI | 2 years after randomisation
  Non-fatal repeat MI requires the presence of two of the following three: symptoms of myocardial ischaemia, a characteristic rise and fall in cardiac markers and a typical ECG pattern involving the development of Q waves or persistent T wave changes.
Heart failure | 2 years after randomisation
  Heart failure is defined as symptoms or signs consistent with congestive heart failure with use of intravenous decongestive therapy greater than 2 hours (IV diuretics, IV nesiritide, IV inotropes) in a patient not requiring hospital admission, or, augmented heart failure regimen with oral or intravenous medications in patients requiring hospital admission.
Inappropriate ICD denial | 2 years after randomisation
  Inappropriate ICD denial will be defined as patients who did not receive an ICD based on their intervention allocation, who went on to have documented non-fatal arrhythmia or sudden cardiac death.
Appropriate ICD activations (in patients with ICD) | 2 years after randomisation
  Appropriate ICD activation will be defined as ventricular tachyarrhythmia due to VT which meets the treatment criteria defined above or VF.
Inappropriate ICD activations (in patients with ICD) | 2 years after randomisation
  Inappropriate ICD activations will include supra-ventricular tachycardia, atrial fibrillation/flutter, T wave over-sensing, sinus tachycardia and noise from lead complications or extraneous noise.
Complications or re-hospitalisation associated with ICD implantation (in patients with ICD) | 2 years after randomisation
  Complications or re-hospitalisation associated with ICD implantation (in patients with ICD)

CONTACTS AND LOCATIONS:
Overall Officials: Study Principal Investigator Study Principal Investigator, Principal Investigator — Western Sydney Local Health District
Locations (52):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States
- Australia (19):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Nepean Hospital, Kingswood, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Carins Hospital, Cairns, Queensland
  - The Prince Charles Hospital, Chermside, Queensland
  - The Townsville Hospital, Douglas, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - MonashHeart, Clayton, Victoria
  - Northern Hospital, Epping, Victoria
  - Austin Hospital, Melbourne, Victoria
  - Western Health, Sunshine and Footscray Hospitals, Melbourne, Victoria
- Institute for Clinical and Experimental Medicine, Prague, Czechia
- Germany (5):
  - Cardiovascular Center Bad Neustadt, Bad Neustadt an der Saale
  - Klinikum Brandenburg, Brandenburg
  - Universitaetsmedizin Gittingen (University of Göttingen Medical Center), Göttingen
  - Leipzig Heart Center, Leipzig
  - Universitätsklinikum Leipzig, Leipzig
- Greece (3):
  - General Hospital of Athens Giorgios Gennimatas, Athens
  - General Hospital of Athens Ippokrateio, Athens
  - University Hospital of Heraklion Crete, Heraklion
- Hungary (3):
  - Semmelweis University Heart and Vascular Center, Budapest
  - University of Debrecen, Debrecen
  - University of Pécs, Pécs
- Sharee Zadek Medical Centre, Jerusalem, Israel
- Paul Stradins University Clinic, Riga, Latvia
- Malaysia (2):
  - Institut Jantung Negara Sdn Bhd, Kuala Lumpur
  - Pusat Jantung Sarawak (PJS)(Sarawak Heart Centre), Kuala Lumpur
- New Zealand (5):
  - Auckland City Hospital, Grafton, Auckland
  - Middlemore Hospital, Otahuhu, Auckland
  - Waikato Hospital, Hamilton W., Hamilton
  - Christchurch Hospital, Christchurch
  - Wellington Hospital, Wellington
- Poland (4):
  - Medical University of Łódź - Biegański Provincial Specialist Hospital, Lodz
  - Medical University of Łódź - WAM Hospital, Lodz
  - Medical University of Łódź, Lodz
  - National Institute of Cardiology Warsaw, Warsaw
- Russia (2):
  - Almazov National Medical Research Centre, Saint Petersburg
  - Samara State Medical University, Samara
- National University Heart Centre, Singapore (NUHCS), Singapore, Singapore
- The National Institute of Cardiovascular Diseases, Bratislava, Slovakia
- Switzerland (3):
  - University Hospital Basel, Basel
  - University Hospital Bern, Bern
  - Lausanne University Hospital, Lausanne